CLINICAL TRIAL: NCT02566993
Title: Phase III Randomized Clinical Trial of Lurbinectedin (PM01183)/Doxorubicin Versus Cyclophosphamide, Doxorubicin and Vincristine (CAV) or Topotecan as Treatment in Patients With Small-Cell Lung Cancer (SCLC) Who Failed One Prior Platinum-containing Line (ATLANTIS)
Brief Title: Clinical Trial of Lurbinectedin (PM01183)/Doxorubicin Versus CAV or Topotecan as Treatment in Patients With Small-Cell Lung Cancer
Acronym: ATLANTIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-C-003-14
Record Dates: First submitted 2015-09-24; First posted 2015-10-02 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-08

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; Doxorubicin; Cyclophosphamide; Vincristine; Topotecan

ARMS (3):
- Experimental Arm (Experimental): Lurbinectedin (PM01183) / Doxorubicin
  Interventions: Drug: Lurbinectedin (PM01183); Drug: Doxorubicin (DOX)
- Control Arm 1 (Active Comparator): CAV (Cyclophosphamide (CTX), Doxorubicin (DOX) and Vincristine (VCR))
  Interventions: Drug: Doxorubicin (DOX); Drug: Cyclophosphamide (CTX); Drug: Vincristine (VCR)
- Control Arm 2 (Active Comparator): Topotecan
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Lurbinectedin (PM01183)
  Arms: Experimental Arm
Drug: Doxorubicin (DOX)
  Arms: Control Arm 1; Experimental Arm
Drug: Cyclophosphamide (CTX)
  Arms: Control Arm 1
Drug: Vincristine (VCR)
  Arms: Control Arm 1
Drug: Topotecan
  Arms: Control Arm 2

SUMMARY:
Phase III randomized clinical trial of lurbinectedin (PM01183)/doxorubicin (DOX) versus cyclophosphamide (CTX), doxorubicin (DOX) and vincristine (VCR) (CAV) or topotecan as treatment in patients with small-cell lung cancer (SCLC) who failed one prior platinum-containing line.

DETAILED DESCRIPTION:
Multicenter, open-label, randomized, controlled phase III clinical trial to evaluate and compare the activity and safety of an experimental arm consisting of PM01183/DOX combination followed by PM01183 alone, if applicable vs. best Investigator's choice between CAV or topotecan as a control arm, in SCLC patients who failed one prior platinum-containing line but no more than one prior chemotherapy-containing line.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent
2. Adult patients ≥ 18 years
3. Histologically or cytologically confirmed diagnosis of limited or extensive stage SCLC which failed one prior platinum-containing regimen and with a chemotherapy-free interval (CTFI, time from the last dose of first-line chemotherapy to the occurrence of progressive disease) ≥ 30 days. Small-cell carcinoma of unknown primary site with or without neuroendocrine features confirmed in histology test(s) performed on metastatic lesion(s) are eligible, if Ki-67/MIB-1 is expressed in >50% of tumor cells.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2.
5. Adequate hematological, renal, metabolic and hepatic function within 7-10 days prior to randomization
6. At least three weeks since last prior anticancer treatment and adequate recovery from prior treatment toxicity
7. Prior radiotherapy (RT): At least four weeks since completion of whole-brain irradiation, at least two weeks since completion of prophylactic cranial irradiation, and to any other site.
8. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure up to six weeks after treatment discontinuation. Fertile male patients with WOCBP partners should use condoms during treatment and for four months following the last investigational medicinal product dose.

Exclusion Criteria:

1. More than one prior chemotherapy-containing line(re-challenge with the same initial regimen is not allowed)
2. Patients who never received platinum-containing regimen for Small-cell Lung Cancer (SCLC)
3. Prior treatment with PM01183, topotecan or anthracyclines.
4. Limited-stage patients who are candidates for local or regional therapy
5. Impending need for palliative RT or surgery for pathological fractures and/or for medullary compression within four weeks prior to randomization.
6. Symptomatic or progressing or steroid requiring Central Nervous System (CNS) involvement disease at least four weeks prior to randomization
7. Concomitant diseases/conditions:

   Angina, myocardial infarction, congestive heart failure or clinically significant valvular heart disease, arrhythmia, immunodeficiency (including known HIV seropositive), ongoing or treatment-requiring chronic liver disease, active infection, oxygen requirement within two weeks prior to randomization, diffuse interstitial lung disease (ILD) or pulmonary fibrosis, second invasive malignancy treated with chemotherapy and/or radiotherapy, invasive fungal infections requiring systemic treatment within 12 weeks of randomization.
8. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (160):
- United States (29):
  - Alabama Oncology, Birmingham, Alabama
  - Ironwood Physicians P.C. dba Ironwood Cancer & Research Centers, Chandler, Arizona
  - St Jude Hospital Yorba Linda dba St Joseph Heritage Healthcare, Fullerton, California
  - Loma Linda University Medica! Center, Loma Linda, California
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - Boca Raton Regional Hospital Lynn Cancer Institute, Boca Raton, Florida
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - East Jefferson Hematology-Oncology Metairie Physicians Services, Inc, Metairie, Louisiana
  - Anne Arundel Medical Center Oncology and Hematology, Annapolis, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - QUEST Research Institute, Royal Oak, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Summit Medical Group, P.A., Florham Park, New Jersey
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Associates in Hematology and Oncology, P.C., Upland, Pennsylvania
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Tyler Hematology-Oncology PA, Tyler, Texas
  - Medical Oncology Associates PS (dba Summit Cancer Centers), Spokane, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (5):
  - Instituto Médico Especializado Alexander Fleming, C.a.b.a., Buenos Aires
  - Centro para la Atención Integral del Paciente Oncológico (CAIPO), San Miguel de Tucumán, Tucumán Province
  - Instituto Oncológico de Córdoba (IONC), Córdoba
  - CORI - Centro Oncológico Riojano Integral, La Rioja
  - ISIS Centro Especializado de Luce S.A., Santa Fe
- Austria (2):
  - Universitätsklinik für Innere Medizin III der PMU, Salzburg
  - Medizinische Universität Wien / AKH Wien, Universitätsklinik für Innere Medizin I, Abteilung für klinische Onkologie, Vienna
- Belgium (6):
  - AZ Maria Middelares, Ghent
  - Clinique André Renard, Herstal
  - CHR de la citadelle, Liège
  - CHU de Liege - Sart Tilman, Liège
  - CHU Ambroise Paré, Mons
  - AZ Delta Campus Wilgenstraat, Roeselare
- Brazil (10):
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - lOP- Instituto de oncologia do paraná, Curitiba, Paraná
  - Coordenação de Pesquisa Clínica / Instituto Nacional de Câncer, Rio de Janeiro, Rio de Janeiro
  - Instituto COl de Pesquisa, Educação e Gestão, Rio de Janeiro, Rio de Janeiro
  - Associação Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - lrmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de clínicas de Porto alegre, Pôrto Alegre, Rio Grande do Sul
  - Fundação PlO XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - lnstituto de Ensino e Pesquisa Säo Lucas - IEP Säo Lucas, São Paulo, São Paulo
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment - Uni Hospital, Panagyurishte, Panagyurishte
  - Multiprofile Hospital for Active Treatment of Women Health - "Nadezhda", Sofia; Clinic of Medical Oncology, Sofia
  - University Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski", Sofia, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment. EOOD, Sofia; Clinic of Medical Oncology, Sofia
- Canada (6):
  - Southlake Regional Health Centre - Stronach Regional Cancer Centre, Newmarket, Ontario
  - R.S. Mc Laughlin Durham Regional Cancer Centre, Lakeridge Health, Oshawa, Ontario
  - Centre intégré de santé et de services sociaux de la Montérégie Centre, Greenfield Park, Quebec
  - Montreal Oncology Research Inc., Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Biron (Clinique René Laennec), Mount Royal, Quebec
- Czechia (2):
  - Vitkovicka nemocnice, a.s., Plicni oddeleni, Ostrava
  - Krajska zdravotni a.s. Masarykova nemocnice o.z., Ústí nad Labem
- France (7):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Lyon Sud - Service de Pneumologie, Lyon
  - Hôpital Nord - Service Oncologie Multidisciplinaire et Innovations Thérapeutiques, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU de Rennes Hôpital Pontchaillou, Rennes
- Germany (20):
  - Central Clinic of Bad Berka, Bad Berka
  - Vivantes Klinikum am Urban, Hämatologie und Onkologie, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Uniklinik Freiburg, Hämatologie, Onkologie & Stammzellransplantation, Freiburg im Breisgau
  - Asklepios-Fachkliniken München Gauting, Gauting
  - Center for Pneumology and Thoracic Surgery, Gerlingen
  - Thoraxklinik Heidelberg GmbH, Heidelberg
  - Lungenklinik Hemer, Hemer
  - VIDIA Christliche Kliniken Karlsruhe, Karlsruhe
  - Katholisches Klinikum Koblenz-Montabaur, Marienhof Koblenz, Koblenz
  - Onkologische Schwerpunktpraxis Leer-Emden, Leer
  - Klinik Löwenstein gGmbH, Med. Klinik II Onkologie, Löwenstein
  - Uniklinikum Mannheim, TTZ, Medizinische Fakultät Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Klinik für Hämatologie, Onkologie und Palliativmedizin, Minden
  - University of Munich LMU, Dpt. of Medicine V, München
  - Städtisches Krankenhaus München Neuperlach, München
  - Klinikum Bogenhausen, Städt. Klinikum München GmbH, Klinik für Pneumologie und Pneumologische Onkologie, München
  - Klinikum Nürnberg Nord - Pneumologische Onkologie, Nuremberg
  - Universitätsklinikum Ulm - Klinik für Innere Medizin II, Pneumologie, Ulm
  - Medizinische Klinik I, Wuppertal
- Greece (4):
  - University General Hospital of Heraklion - General Hospital "Venizeleio", Heraklion, Crete
  - General Hospital of Chest Diseases of Athens "Sotiria", Athens
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", 2nd Internal Medicine-Oncology Clinic, Athens
  - General Hospital of Thessaloniki "G. Papanikolaou", Pulmonary Clinic, Aristotle University of Thessaloniki, Thessaloniki
- Hungary (9):
  - Országos Korányi TBC és Pulmonológiai Intézet, 6. Pulmonológia és Bronchologia, Budapest
  - Országos Korányi TBC és Pulmonológiai lntézet, 14. Pulmonológia, Budapest
  - Veszprém Megyei Tüdögyógyintézet, 3. Pulmonológiai Osztály, Farkasgyepű
  - Mátrai Gyógyintézet, Bronchológia, Mátraháza
  - Miskolci Semmelweis Kórház és Egyetemi Oktatókórház, Pulmonológiai Osztály, Miskolc
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, I. Pulmonológiai Osztály, Székesfehérvár
  - Markusovszky Egyetemi Oktatókórház, Pulmonológiai Osztály, Szombathely
  - Szent Borbála Kórház, Pulmonológiai osztály, Tatabánya
  - Zala Megyei Kórház, Pulmonologia, Zalaegerszeg
- Italy (9):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - IRCCS CROB (Istituto di Ricovero e Cura a Carattere Scientifico), Rionero in Vulture, PZ
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Azienda Ospedaliero - Universitaria "Policlinico - Vittorio Emanuele" - Presidio G. Rodolico, Catania
  - AOU Maggiore della Carità - SC Oncologia, Novara
  - Istituto Oncologico Veneto, Padua
  - lRCCS-Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - ASST della Valtellina e dell' Alto Lario P.O. Di Sondrio, Sondrio
- Lebanon (5):
  - Ain Wazein Hospital, Ain Wazein, El Chouf
  - American University of Beirut Medical Center, Beirut
  - Hotel Dieu de France, Beirut
  - Centre Hospitalier Universitaire Notre Dame de Secours, Byblos
  - Hammoud Hospital University Medical Center, Sidon
- Netherlands (4):
  - The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Spaarne Gasthuis, Hoofddorp
  - MUMC, Maastricht
  - Maxima Medisch Centrum, Veldhoven
- Poland (4):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie; Oddzial Onkologii Klinicznej im. dr Ewy Pileckiej z pododdzialem, Bialystok
  - Szpitale Pomorskie Sp. z o.o., Oddzial Onkologii Klinicznej, Oddzial Onkologii i Radioterapii, Gdynia
  - Mazowieckie Centrum Leczenia Chorób Pluc i Gruźlicy Oddzial III Chorób Pluc z Pododdzialem Onkologicznym, Otwock
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. K.Marcinkowskiego w Poznaniu, Oddzial Chemioterapii, Poznan
- Portugal (6):
  - Centro Clínico Champalimaud - Fundação Champalimaud, Lisbon
  - Centro Hospitalar Lisboa Norte, EPE- Hospital Pulido Valente, Lisbon
  - Centro Hospitalar do Porto, EPE - Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de São João, EPE, Porto
- Romania (7):
  - SC Centrul de Oncologie Sf. Nectarie SRL, Departament Oncologie Medícala, Craiova, Dolj
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei", Constanța, Judet Constanta
  - SC Oncolab SRL, Craiova, Judet Dolj
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris", Sectia Oncologie Medicala, Baia Mare, Maramureş
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj-Napoca, Departament Oncologie Medicala, Cluj-Napoca
  - Institutul Oncologic "Prof. Dr. lon Chiricuta" Cluj-Napoca, Dcpartamentul Oncologie Medicala, Cluj-Napoca
  - Institutul Oncologic "Prof. Dr. lon Chiricuta" Cluj-Napoca, Sectia Oncologic Medicala, Cluj-Napoca
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol ICO, Badalona, Barcelona
  - Corporació Sanitaria Parc Taulí-Hospital de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo hospitalario regional virgen rocío, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - The Christie NHS Fundation Trust, Manchester, Greater Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Bristol Cancer Institute, UHB NHS Foundation Trust, Bristol
  - University College London Hospitals NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK, London
  - Worcestershire Acute Hospitals NHS Trust, Worcester

REFERENCES:
- [Derived] Aix SP, Ciuleanu TE, Navarro A, Cousin S, Bonanno L, Smit EF, Chiappori A, Olmedo ME, Horvath I, Grohe C, Farago AF, Lopez-Vilarino JA, Cullell-Young M, Nieto A, Vasco N, Gomez J, Kahatt C, Zeaiter A, Carcereny E, Roubec J, Syrigos K, Lo G, Barneto I, Pope A, Sanchez A, Kattan J, Zarogoulidis K, Waller CF, Bischoff H, Juan-Vidal O, Reinmuth N, Domine M, Paz-Ares L. Combination lurbinectedin and doxorubicin versus physician's choice of chemotherapy in patients with relapsed small-cell lung cancer (ATLANTIS): a multicentre, randomised, open-label, phase 3 trial. Lancet Respir Med. 2023 Jan;11(1):74-86. doi: 10.1016/S2213-2600(22)00309-5. Epub 2022 Oct 14. PMID 36252599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first randomization took place on 30 August 2016 and the first study treatment was administered on 25 October 2016. The cutoff date for results presented in this Clinical Study Report was 24 February 2020.
  A total of 919 patients were screened; 613 of these 919 patients were randomized at a 1:1 ratio to receive any of the study treatments at 135 investigational sites from 20 countries.
Groups:
- Lurbinectedin/Doxorubicin: Doxorubicin: 40.0 mg/m2 i.v. on Day 1 through peripheral or central lines (according to local label), followed by, Lurbinectedin: 2.0 mg/m2 i.v. as a 1-hour infusion on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines. A minimum volume of 100 mL diluted in 5% glucose or 0.9% sodium chloride solution for infusion, had to be used for administration through a central venous catheter; if a peripheral venous catheter was used, the minimum volume was 250 mL.
  The combination was to be administered for up to a maximum of ten cycles.
- Topotecan or Cyclophosphamide/Doxorubicin/Vincristine: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and Cyclophosphamide, Doxorubicin and Vincristine (CAV), until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  Topotecan: i.v. daily on Days 1-5 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines (according to local label) at the following doses:
  * 1.50 mg/m2 daily, for patients with calculated Creatinine Clearance (CrCL) ≥60 mL/min.
  * 1.25 mg/m2 daily, for patients with calculated CrCL between 40 and 59 mL/min.
  * 0.75 mg/m2 daily, for patients with calculated CrCL between 30 and 39 mL/min.
  or
  CAV: i.v. on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines at the following doses:
  * Cyclophosphamide: 1000 mg/m2,
  * Doxorubicin: 45.0 mg/m2,
  * Vincristine: 2.0 mg flat dose. The triple combination was to be administered for up to a maximum of ten cycles
Period: Overall Study
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Started | 307 | 306
Completed | 0 | 0
Not Completed | 307 | 306
Not completed — Randomized but not treated | 5 | 16
Not completed — Progressive disease | 213 | 152
Not completed — Withdrawal by Subject | 12 | 28
Not completed — Death | 17 | 23
Not completed — Physician Decision | 10 | 17
Not completed — Study drug-related adverse event | 20 | 41
Not completed — Non study drug-related adverse event | 9 | 9
Not completed — Symptomatic deterioration | 9 | 16
Not completed — End of study due to events required for OS analysis according to study protocol had been reached | 9 | 1
Not completed — Sponsor's decision after incorrect treatment at site | 1 | 1
Not completed — Screening failure | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Symptomatic deterioration, progression disease, and a decision by the Investigator | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Topotecan or Cyclophosphamide/Doxorubicin/Vincristine: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and CAV, until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  Topotecan: i.v. daily on Days 1-5 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines (according to local label) at the following doses:
  * 1.50 mg/m2 daily, for patients with calculated CrCL ≥60 mL/min.
  * 1.25 mg/m2 daily, for patients with calculated CrCL between 40 and 59 mL/min.
  * 0.75 mg/m2 daily, for patients with calculated CrCL between 30 and 39 mL/min.
  or
  CAV: i.v. on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines at the following doses:
  * Cyclophosphamide: 1000 mg/m2,
  * Doxorubicin: 45.0 mg/m2,
  * Vincristine: 2.0 mg flat dose. The triple combination was to be administered for up to a maximum of ten cycles
- Total: Total of all reporting groups
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine | Total
Number analyzed (Participants) | 307 | 306 | 613
Age, Continuous [Median (Full Range); unit: years] | 63.0 [19 to 83] | 63.0 [37 to 82] | 63 [19 to 83]
Age, Customized [Count of Participants; unit: Participants]
  18-49 years | 16 | 13 | 29
  50-65 years | 161 | 166 | 327
  >65 years | 130 | 127 | 257
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 133 | 264
  Male | 176 | 173 | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 266 | 265 | 531
  Black or African American | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Other | 2 | 2 | 4
  Not available | 38 | 37 | 75
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 3 | 4 | 7
  Romania | 20 | 19 | 39
  Hungary | 23 | 23 | 46
  United States | 32 | 30 | 62
  Czechia | 4 | 5 | 9
  United Kingdom | 10 | 11 | 21
  Portugal | 10 | 5 | 15
  Spain | 62 | 63 | 125
  Greece | 12 | 13 | 25
  Lebanon | 8 | 9 | 17
  Canada | 10 | 7 | 17
  Austria | 5 | 3 | 8
  Netherlands | 9 | 9 | 18
  Belgium | 9 | 12 | 21
  Brazil | 13 | 15 | 28
  Poland | 7 | 6 | 13
  Italy | 21 | 20 | 41
  Bulgaria | 5 | 6 | 11
  France | 11 | 12 | 23
  Germany | 33 | 34 | 67
Weight [Median (Full Range); unit: Kg] | 73.0 [40 to 143] | 74.0 [38 to 158] | 73.4 [37.9 to 158]
Height [Median (Full Range); unit: cm] | 168 [145 to 196] | 168 [146 to 191] | 168 [145 to 196]
Body surface area [Median (Full Range); unit: m^2] | 1.8 [1.4 to 2.5] | 1.8 [1.3 to 2.8] | 1.8 [1.3 to 2.8]
Body mass index [Median (Full Range); unit: Kg/m^2] | 25.9 [15.3 to 51.2] | 26.0 [14.8 to 43.8] | 25.9 [14.8 to 51.2]
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status (ECOG PS) PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 95 | 95 | 190
    PS 1 | 197 | 204 | 401
    PS 2 | 15 | 7 | 22
Smoking status [Count of Participants; unit: Participants]
  Former | 197 | 199 | 396
  Current | 91 | 89 | 180
  Never | 19 | 18 | 37
Time from first diagnosis to randomization [Median (Full Range); unit: months] | 9.3 [2.5 to 55.5] | 9.1 [2.3 to 42.3] | 9.2 [2.5 to 55.5]
Disease stage [Count of Participants; unit: Participants] — Limited stage. Limited stage means that the cancer is only in 1 part of the chest and radiation therapy could be a treatment option.
  Extensive stage. Extensive stage is used to describe SCLC that has spread to other parts of the body such as the opposite lung, bone, brain, or bone marrow.
  Participants
    Limited | 25 | 28 | 53
    Extensive | 282 | 278 | 560
Number of sites involved [Count of Participants; unit: Participants]
  <3 sites | 38 | 31 | 69
  ≥3 sites | 269 | 275 | 544
Number of sites involved [Median (Full Range); unit: sites] | 4.0 [1 to 10] | 4.0 [2 to 11] | 4.0 [1 to 11]
Bulky disease [Count of Participants; unit: Participants] — Bulky disease defined as one lesion ≥50 mm
  Participants | 144 | 127 | 271
Central Nervous System involvement [Count of Participants; unit: Participants] | 46 | 49 | 95
Paraneoplastic syndrome [Count of Participants; unit: Participants] | 9 | 11 | 20
Prior radiotherapy [Count of Participants; unit: Participants] | 237 | 236 | 473
Prior surgery [Count of Participants; unit: Participants] | 27 | 39 | 66
Lines of anticancer therapy [Median (Full Range); unit: lines of therapies] | 1.0 [1 to 2] | 1.0 [1 to 2] | 1.0 [1 to 2]
Best response to last prior chemotherapy [Count of Participants; unit: Participants] — Complete response (CR): disappearance of all lesions; Partial response (PR): ≥10% decrease in target lesion size or ≥15% decrease in tumor density; Disease progression (PD): ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; Stable disease (SD): none of the CR, PR, or PD criteria met; Unknown (UK)
  Participants
    Complete response | 17 | 15 | 32
    Partial response | 192 | 191 | 383
    Stable disease | 71 | 63 | 134
    Progressive disease | 17 | 21 | 38
    Unknown | 10 | 16 | 26
Prior immunotherapy against PD-1 or PD-L1 [Count of Participants; unit: Participants] — PD-1, programmed cell death protein-1; PD-L1, programmed death ligand-1
  Participants | 19 | 17 | 36
Time-to-progression to prior chemotherapy [Median (Full Range); unit: months] | 7.4 [0.8 to 40.2] | 7.4 [1.6 to 33.7] | 7.4 [0.8 to 40.2]
Time from last prior progressive disease to randomization [Median (Full Range); unit: days] | 25.0 [3 to 621] | 25.5 [1 to 327] | 25.0 [1.0 to 621]
Time from end date of last prior chemotherapy to randomization [Median (Full Range); unit: days] | 157.0 [28.0 to 1545.0] | 153.0 [29.0 to 1151.0] | 155 [28 to 1545]
Chemotherapy-free interval [Median (Full Range); unit: days] | 115.0 [0 to 1094] | 120.5 [13 to 960] | 120 [0 to 1094]
Chemotherapy-free interval [Count of Participants; unit: Participants]
  <90 days | 99 | 101 | 200
  90-179 days | 115 | 116 | 231
  ≥180 days | 93 | 89 | 182

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be calculated from the date of randomization to the date of death (death event) or last contact(in this case, survival will be censored on that date).
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Topotecan or Cyclophosphamide/Doxorubicin/Vincristine: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and CAV, until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  Topotecan: i.v. daily on Days 1-5 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines (according to local label) at the following doses:
  * 1.50 mg/m2 daily, for patients with calculated CrCL ≥60 mL/min.
  * 1.25 mg/m2 daily, for patients with calculated CrCL between 40 and 59 mL/min.
  * 0.75 mg/m2 daily, for patients with calculated CrCL between 30 and 39 mL/min.
  or
  CAV: i.v. on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines at the following doses:
  * Cyclophosphamide: 1000 mg/m2,
  * Doxorubicin: 45.0 mg/m2,
  * Vincristine: 2.0 mg flat dose (FD). The triple combination was to be administered for up to a maximum of ten cycles
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
months | 8.6 [7.1 to 9.4] | 7.6 [6.6 to 8.2]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.9029, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 0.967, 95% CI 2-sided [0.815 to 1.148]

2. Secondary Outcome: Difference in Overall Survival Between Lurbinectedin/Doxorubicin (DOX) and CAV in Patients With CAV as Best Investigator's Choice: Overall Survival Rate at 12 Months
Description: as for outcome 1
Time Frame: At 12 months
Population: Patients with Cyclophosphamide, Doxorubicin and Vincristine (CAV) as best Investigator's choice
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Topotecan or Cyclophosphamide/Doxorubicin/Vincristine: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and CAV, until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  Topotecan: i.v. daily on Days 1-5 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines (according to local label) at the following doses:
  * 1.50 mg/m2 daily, for patients with calculated CrCL ≥60 mL/min.
  * 1.25 mg/m2 daily, for patients with calculated CrCL between 40 and 59 mL/min.
  * 0.75 mg/m2 daily, for patients with calculated CrCL between 30 and 39 mL/min.
  or
  CAV: i.v. on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines at the following doses:
  * Cyclophosphamide: 1000 mg/m2,
  * Doxorubicin: 45.0 mg/m2,
  * Vincristine: 2.0 mg FD. The triple combination was to be administered for up to a maximum of ten cycles
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 184 | 179
percentage of participants | 29.6 [22.8 to 36.3] | 24.4 [17.9 to 31.0]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.2826, Normal test

3. Secondary Outcome: Difference in Overall Survival Between Lurbinectedin/DOX and CAV in Patients With CAV as Best Investigator's Choice: Overall Survival Rate at 18 Months
Description: as for outcome 1
Time Frame: At 18 months
Population: Patients with Cyclophosphamide, Doxorubicin and Vincristine (CAV) as best Investigator's choice
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 184 | 179
percentage of participants | 13.9 [8.8 to 19.1] | 15.9 [10.3 to 21.4]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.6216, Normal test

4. Secondary Outcome: Difference in Overall Survival Between Lurbinectedin/DOX and CAV in Patients With CAV as Best Investigator's Choice: Overall Survival Rate at 24 Months
Description: as for outcome 1
Time Frame: At 24 months
Population: Patients with Cyclophosphamide, Doxorubicin and Vincristine (CAV) as best Investigator's choice
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 184 | 179
percentage of participants | 8.6 [4.1 to 13.1] | 8.7 [4.1 to 13.4]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.9708, Normal test

5. Secondary Outcome: Progression-free Survival (PFS) by Independent Review Committee
Description: Progression-free survival (PFS) is defined as the time from the date of randomization to the date of documented progression per RECIST v.1.1 or death (regardless of the cause of death). If the patient receives further antitumor therapy or is lost to follow-up before PD, PFS will be censored at the date of last tumor assessment before the date of subsequent antitumor therapy.
Time Frame: Every six weeks up to progression disease, a period of approximately 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
months | 4.0 [2.8 to 4.2] | 4.0 [3.0 to 4.1]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.3257, Log Rank; Stratified log-rank test; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.693 to 0.996]

6. Secondary Outcome: Progression-free Survival Rate at 6 Months by Independent Review Committee
Description: as for outcome 5
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
percentage of participants | 31.3 [25.7 to 36.8] | 24.4 [18.9 to 29.9]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.0851, Normal test

7. Secondary Outcome: Progression-free Survival Rate at 12 Months by Independent Review Committee
Description: as for outcome 5
Time Frame: at 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
percentage of participants | 10.8 [6.7 to 14.9] | 4.4 [1.4 to 7.4]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.0129, Normal test

8. Secondary Outcome: Best Antitumor Response by Independent Review Committee
Description: Best antitumor response will be the best response obtained in any evaluation according to RECIST v.1.1.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; UK,unknown
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
Participants
  Complete response | 8 | 4
  Partial response | 89 | 87
  Stable disease | 111 | 116
  Progressive disease | 74 | 52
  Unknown | 25 | 47

9. Secondary Outcome: Overall Response Rate by Independent Review Committee
Description: Overall response rate is defined as the proportion of patients who have a partial or complete response in the best antitumor response. The best antitumor response will be the best response obtained in any evaluation according to RECIST v.1.1.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; UK,unknown
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 307 | 306
percentage of participants | 31.6 [26.4 to 37.1] | 29.7 [24.7 to 35.2]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.6616, Binomial test

10. Secondary Outcome: Duration of Response by Independent Review Committee
Description: Duration of Response is defined as the time that patients who have a partial or complete response in the best antitumor response. The best antitumor response will be the best response obtained in any evaluation according to RECIST v.1.1.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; UK,unknown
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: Patients who have a partial or complete response in the best antitumor response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 97 | 91
months | 5.7 [4.1 to 7.1] | 3.8 [2.8 to 4.3]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; p = 0.0012, Log Rank; Hazard Ratio (HR) = 0.581, 95% CI 2-sided [0.416 to 0.812]

11. Secondary Outcome: Overall Survival in Patients With Chemotherapy-free Interval ≥ 90 Days
Description: as for outcome 1
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: A preplanned exploratory efficacy subgroup analysis was focused on patients had chemotherapy-free interval ≥90 days after first-line chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 208 | 205
months | 10.3 [9.0 to 11.8] | 8.7 [7.8 to 9.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.744 to 1.140]

12. Secondary Outcome: Progression-free Survival in Patients With Chemotherapy-free Interval ≥90 Days
Description: as for outcome 5
Time Frame: Every six weeks up to progression disease, a period of approximately 3.5 years
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 208 | 205
months | 4.8 [4.1 to 5.6] | 4.4 [4.0 to 5.3]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.688, 95% CI 2-sided [0.549 to 0.863]

13. Secondary Outcome: Best Antitumor Response in Patients With Chemotherapy-free Interval ≥ 90 Days
Description: as for outcome 8
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 208 | 205
Participants
  Complete response | 8 | 4
  Partial response | 69 | 68
  Stable disease | 85 | 73
  Progression disease | 32 | 35
  Unknown | 14 | 25

14. Secondary Outcome: Overall Response Rate in Patients With Chemotherapy-free Interval ≥ 90 Days
Description: as for outcome 9
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 208 | 205
percentage of participants | 37.0 [30.4 to 44.0] | 35.1 [28.6 to 42.1]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.616 to 1.376]

15. Secondary Outcome: Duration of Response in Patients With Chemotherapy-free Interval ≥ 90 Days
Description: as for outcome 10
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: Patients who have a partial or complete response in the best antitumor response. A preplanned exploratory efficacy subgroup analysis was focused on patients had chemotherapy-free interval ≥90 days after first-line chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 77 | 72
months | 6.9 [4.1 to 8.3] | 4.0 [3.0 to 4.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.504, 95% CI 2-sided [0.346 to 0.736]

16. Secondary Outcome: Overall Survival in Patients With Chemotherapy-free Interval < 90 Days
Description: as for outcome 1
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: A preplanned exploratory efficacy subgroup analysis was focused on patients had chemotherapy-free interval <90 days after first-line chemotherapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 99 | 101
months | 5.7 [4.1 to 6.7] | 5.3 [4.2 to 6.1]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.122, 95% CI 2-sided [0.840 to 1.500]

17. Secondary Outcome: Progression-free Survival in Patients With Chemotherapy-free Interval <90 Days
Description: as for outcome 5
Time Frame: Every six weeks up to progression disease, a period of approximately 3.5 years
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 99 | 101
months | 1.6 [1.4 to 2.7] | 2.8 [2.5 to 3.0]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.306, 95% CI 2-sided [0.955 to 1.786]

18. Secondary Outcome: Best Antitumor Response in Patients With Chemotherapy-free Interval <90 Days
Description: as for outcome 8
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 99 | 101
Participants
  Partial response | 20 | 19
  Stable disease | 26 | 43
  Progression disease | 42 | 17
  Unknown | 11 | 22

19. Secondary Outcome: Overall Response Rate in Patients With Chemotherapy-free Interval <90 Days
Description: as for outcome 9
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 99 | 101
percentage of participants | 20.2 [12.8 to 29.5] | 18.8 [11.7 to 27.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.915, 95% CI 2-sided [0.455 to 1.843]

20. Secondary Outcome: Duration of Response in Patients With Chemotherapy-free Interval <90 Days
Description: as for outcome 10
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: Patients who have a partial or complete response in the best antitumor response. A preplanned exploratory efficacy subgroup analysis was focused on patients had chemotherapy-free interval <90 days after first-line chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 20 | 19
months | 3.0 [1.4 to 4.5] | 2.8 [1.4 to 4.1]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.092, 95% CI 2-sided [0.506 to 2.360]

21. Secondary Outcome: Overall Survival in Patients Without Central Nervous System Involvement at Baseline
Description: as for outcome 1
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: A preplanned exploratory efficacy subgroup analysis was focused on patients without Central Nervous System Involvement at Baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 261 | 257
months | 9.1 [8.1 to 10.2] | 7.7 [6.7 to 8.6]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.765 to 1.113]

22. Secondary Outcome: Progression-free Survival in Patients Without Central Nervous System Involvement at Baseline
Description: as for outcome 5
Time Frame: Every six weeks up to progression disease, a period of approximately 3.5 years
Population: as for outcome 21
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 261 | 257
months | 4.2 [3.7 to 4.8] | 4.1 [3.1 to 4.3]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.645 to 0.961]

23. Secondary Outcome: Best Antitumor Response in Patients Without Central Nervous System Involvement at Baseline
Description: as for outcome 8
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 261 | 257
Participants
  Complete response | 7 | 3
  Partial response | 79 | 76
  Stable disease | 101 | 100
  Progression disease | 55 | 40
  Unknown | 19 | 38

24. Secondary Outcome: Overall Response Rate in Patients Without Central Nervous System Involvement at Baseline
Description: as for outcome 9
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 261 | 257
percentage of participants | 33.0 [27.3 to 39.0] | 30.7 [25.2 to 36.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.903, 95% CI 2-sided [0.624 to 1.307]

25. Secondary Outcome: Duration of Response in Patients Without Central Nervous System Involvement at Baseline
Description: as for outcome 10
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: Patients who have a partial or complete response in the best antitumor response. A preplanned exploratory efficacy subgroup analysis was focused on patients without Central Nervous System Involvement at Baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 86 | 79
months | 5.7 [4.1 to 7.3] | 4.0 [3.0 to 4.9]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 0.560, 95% CI 2-sided [0.392 to 0.799]

26. Secondary Outcome: Overall Survival in Patients With Central Nervous System Involvement at Baseline
Description: as for outcome 1
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: A preplanned exploratory efficacy subgroup analysis was focused on patients with Central Nervous System Involvement at Baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 46 | 49
months | 4.6 [3.1 to 6.1] | 6.6 [4.0 to 8.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.291, 95% CI 2-sided [0.838 to 1.990]

27. Secondary Outcome: Progression-free Survival in Patients With Central Nervous System Involvement at Baseline
Description: as for outcome 5
Time Frame: Every six weeks up to progression disease, a period of approximately 3.5 years
Population: as for outcome 26
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 46 | 49
months | 1.9 [1.4 to 2.7] | 2.8 [1.4 to 3.8]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.290, 95% CI 2-sided [0.824 to 2.019]

28. Secondary Outcome: Best Antitumor Response in Patients With Central Nervous System Involvement at Baseline
Description: as for outcome 8
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 46 | 49
Participants
  Complete response | 1 | 1
  Partial response | 10 | 11
  Stable disease | 10 | 16
  Progression disease | 19 | 12
  Unknown | 6 | 9

29. Secondary Outcome: Overall Response Rate in Patients With Central Nervous System Involvement at Baseline
Description: as for outcome 9
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 46 | 49
percentage of participants | 23.9 [12.6 to 38.8] | 24.5 [13.3 to 38.9]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.032, 95% CI 2-sided [0.403 to 2.641]

30. Secondary Outcome: Duration of Response in Patients With Central Nervous System Involvement at Baseline
Description: as for outcome 10
Time Frame: Every three months up to death or study termination, a period of approximately 3.5 years
Population: Patients who have a partial or complete response in the best antitumor response. A preplanned exploratory efficacy subgroup analysis was focused on patients with Central Nervous System Involvement at Baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan or Cyclophosphamide/Doxorubicin/Vincristine
Number analyzed (Participants) | 11 | 12
months | 1.5 [0.1 to NA] — Not reached | 2.7 [1.3 to 4.0]
Statistical Analysis 1: Comparison: Lurbinectedin/Doxorubicin vs Topotecan or Cyclophosphamide/Doxorubicin/Vincristine; Test type: Superiority; Hazard Ratio (HR) = 1.013, 95% CI 2-sided [0.373 to 2.750]

ADVERSE EVENTS:
Time Frame: Patients were assessed through study completion, approximately 2 years
Description: 21 of 613 randomized patients did not receive the study treatment. Safety population consisted of 592 treated patients. 302 had been randomized to lurbinectedin/DOX and 290 to topotecan or CAV. However, one patient randomized to receive topotecan was treated with lurbinectedin/DOX instead. For safety data analysis, this patient has been moved to the lurbinectedin/DOX Arm, and the safety population thereby comprised 303 patients with lurbinectedin/DOX and 289 patients with topotecan or CAV.
Groups:
- Topotecan: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and CAV, until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  Topotecan: i.v. daily on Days 1-5 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines (according to local label) at the following doses:
  * 1.50 mg/m2 daily, for patients with calculated CrCL ≥60 mL/min.
  * 1.25 mg/m2 daily, for patients with calculated CrCL between 40 and 59 mL/min.
  * 0.75 mg/m2 daily, for patients with calculated CrCL between 30 and 39 mL/min.
- Cyclophosphamide/Doxorubicin/Vincristine: If the patient was randomized to the Control Arm, the assigned treatment was based on the reported Investigator's preference between topotecan and CAV, until the first of these options had reached 55% of the target patient enrollment in this arm. Once this had occurred, patients in the Control Arm were to receive the other option.
  CAV: i.v. on Day 1 q3wk (three weeks ±48h = one treatment cycle) through peripheral or central lines at the following doses:
  * Cyclophosphamide: 1000 mg/m2,
  * Doxorubicin: 45.0 mg/m2,
  * Vincristine: 2.0 mg FD. The triple combination was to be administered for up to a maximum of ten cycles
Arm/Group | Lurbinectedin/Doxorubicin | Topotecan | Cyclophosphamide/Doxorubicin/Vincristine
All-Cause Mortality (participants affected / at risk) | 264/303 | 100/121 | 148/168
Serious Adverse Events (participants affected / at risk) | 126/303 | 66/121 | 75/168
Other Adverse Events (participants affected / at risk) | 292/303 | 120/121 | 148/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin/Doxorubicin (N=303) | Topotecan (N=121) | Cyclophosphamide/Doxorubicin/Vincristine (N=168)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 13 (16) | 9 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12) | 7 (8) | 17 (17)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 9 (10) | 12 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (16) | 15 (33) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 5 (5) | 2 (2)
General physical health deterioration (General disorders) | 7 (8) | 4 (5) | 5 (6)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 1 (2) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 5 (6) | 6 (6)
Pneumonia (Infections and infestations) | 14 (18) | 5 (5) | 7 (7)
Sepsis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (11) | 3 (5) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Central pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 2 (5) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurbinectedin/Doxorubicin (N=303) | Topotecan (N=121) | Cyclophosphamide/Doxorubicin/Vincristine (N=168)
Anaemia (Blood and lymphatic system disorders) | 121 (341) | 84 (283) | 89 (250)
Leukopenia (Blood and lymphatic system disorders) | 28 (106) | 32 (77) | 46 (123)
Lymphopenia (Blood and lymphatic system disorders) | 15 (51) | 10 (21) | 13 (61)
Neutropenia (Blood and lymphatic system disorders) | 101 (316) | 74 (173) | 107 (251)
Thrombocytopenia (Blood and lymphatic system disorders) | 70 (246) | 71 (251) | 61 (155)
Abdominal pain (Gastrointestinal disorders) | 14 (17) | 12 (16) | 12 (13)
Constipation (Gastrointestinal disorders) | 59 (90) | 30 (45) | 25 (31)
Diarrhoea (Gastrointestinal disorders) | 43 (65) | 25 (30) | 23 (29)
Nausea (Gastrointestinal disorders) | 123 (219) | 33 (42) | 55 (76)
Vomiting (Gastrointestinal disorders) | 72 (125) | 15 (17) | 33 (36)
Fatigue (General disorders) | 164 (365) | 64 (162) | 79 (152)
Mucosal inflammation (General disorders) | 30 (50) | 5 (7) | 14 (24)
Non-cardiac chest pain (General disorders) | 26 (27) | 7 (9) | 13 (16)
Oedema (General disorders) | 21 (24) | 13 (14) | 7 (7)
Pyrexia (General disorders) | 28 (32) | 12 (19) | 21 (28)
Lower respiratory tract infection (Infections and infestations) | 18 (24) | 10 (15) | 11 (14)
Pharyngitis (Infections and infestations) | 19 (26) | 7 (7) | 5 (6)
Pneumonia (Infections and infestations) | 10 (12) | 6 (6) | 9 (9)
Ejection fraction decreased (Investigations) | 16 (17) | 0 (0) | 9 (11)
Weight decreased (Investigations) | 64 (79) | 14 (19) | 24 (25)
Decreased appetite (Metabolism and nutrition disorders) | 85 (129) | 20 (27) | 40 (61)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (41) | 13 (25) | 12 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (25) | 7 (12) | 14 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 5 (6) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (49) | 13 (19) | 20 (24)
Dizziness (Nervous system disorders) | 28 (31) | 10 (11) | 13 (15)
Headache (Nervous system disorders) | 30 (33) | 13 (14) | 19 (19)
Insomnia (Psychiatric disorders) | 13 (13) | 8 (11) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (80) | 23 (28) | 26 (31)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 (63) | 24 (26) | 24 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 34 (40) | 9 (9) | 27 (36)
Hypotension (Vascular disorders) | 19 (25) | 4 (4) | 13 (14)
General physical health deterioration (General disorders) | 6 (7) | 4 (4) | 9 (9)
Candida infection (Infections and infestations) | 10 (11) | 3 (3) | 11 (12)
Urinary tract infection (Infections and infestations) | 15 (17) | 3 (3) | 10 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (12) | 7 (12) | 6 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14) | 5 (5) | 9 (12)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 4 (4) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02566993/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02566993/SAP_001.pdf